CLINICAL TRIAL: NCT05941858
Title: A Tai Chi Intervention to Promote Smoking Cessation Among Cancer Survivors
Brief Title: Online Tai Chi Intervention to Promote Smoking Cessation Among Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OSU-22271; NCI-2023-04163 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-06-02; First posted 2023-07-12 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: Smoking Cessation; Tai Chi
MeSH Terms: conditions — Neoplasms; Smoking Cessation | interventions — Smoking Devices; Carbon Monoxide; Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study staff conducting data management and analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Tai Chi) (Experimental): Participants receive access to the online WaQi program to practice Tai Chi supervised over 60 minutes BIW and home-based over 10 minutes five days a week for 8 weeks. Participants also receive a document highlighting NCI resources for quitting smoking including NCI's tollfree Quitline number, state Quitline numbers and other resources, and undergo CO testing on study.
  Interventions: Behavioral: Smoking Cessation Intervention; Procedure: Carbon Monoxide Measurement; Other: Internet-Based Intervention; Other: Survey Administration; Other: Tai Chi
- Arm II (Standard cessation) (Active Comparator): Participants receive a document highlighting NCI resources for quitting smoking including NCI's tollfree Quitline number, state Quitline numbers and other resources, and undergo CO testing on study. Participants also receive an 8-week online Tai Chi self-administered teaching module subscription at the end of the study.
  Interventions: Behavioral: Smoking Cessation Intervention; Procedure: Carbon Monoxide Measurement; Other: Internet-Based Intervention; Other: Survey Administration; Other: Tai Chi

INTERVENTIONS:
Behavioral: Smoking Cessation Intervention — Receive smoking cessation resource document
  Other Names: Smoking and Tobacco Use Cessation Interventions
Procedure: Carbon Monoxide Measurement — Undergo CO test
  Other Names: Carbon Monoxide; iCOquit
Other: Internet-Based Intervention — Receive access to WaQi/Tai Chi program
Other: Survey Administration — Ancillary studies
Other: Tai Chi — Practice Tai Chi

SUMMARY:
This clinical trial evaluates an online Tai Chi intervention to promote smoking cessation among cancer survivors. Tai chi is a practice that involves a series of slow gentle movements and physical postures, a meditative state of mind, and controlled breathing. It is a gentle form of exercise that can be done while sitting or standing and does not involve any medications or medical procedures. Tai chi originated as an ancient martial art in China. Over the years, it has become more focused on health promotion and rehabilitation. The use of Tai Chi may be beneficial for cancer patients who want to quit smoking.

DETAILED DESCRIPTION:
Aim 1: The primary objective of this study is to pilot an online Tai Chi intervention promoting smoking cessation among cancer survivors1.

Aim 2: Examine whether an online Tai Chi intervention reduces cigarette dependence among cancer survivors who are aged 21 and are interested in quitting smoking.

Aim 3: Test whether an online Tai Chi intervention increases quit attempts and cessation abstinence among cancer survivors who are aged 21 or older and are interested in quitting smoking.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants participate in an 8-week supervised online WaQi/Tai Chi program. Participants receive standard cessation treatment which includes receiving a document highlighting smoking cessation resources.

ARM II: Participants receive standard cessation treatment which includes receiving a document highlighting smoking cessation resources. Participants also receive an 8-week online Tai Chi self-administered teaching module subscription at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivor (i.e., have had a cancer diagnosis)
* Age 21 years and older
* English speaking/reading
* Report smoking tobacco in the past 30 days
* Report at least moderate interest in quitting smoking (>= 3 on a Likert type scale with 5 being very extremely interested)
* Can participate in Zoom calls for orientation and intervention
* Have access to a smartphone or tablet
* Willing to download a free application (app)
* Can commit to the 8-weeks intervention (WaQi program)
* Are not currently or have not regularly practiced Tai Chi in the last 6 months
* Willing to blow into a device (for carbon monoxide measurements)

Exclusion Criteria:

* Non-cancer survivors
* Patients under 21 years old
* Non-English speaking/reading
* Non-smokers in the past 30 days
* Report lower than moderate interest in quitting smoking (< 3 on a Likert type scale with 5 being very extremely interested)
* Cannot to participate Zoom calls for orientation and intervention
* No access to a smartphone or tablet
* Not willing to download a free app
* Cannot commit to the intervention
* Has practiced Tai Chi regularly in the last 6 months
* Not willing to blow into a device
* Eligible, but sampling quotas full

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation | At baseline, 4 weeks after start of intervention, and 1 week, 3 months and 6 months post-intervention
  Will be assessed by the participants in both groups by carbon monoxide (CO) verification and self-administered online surveys.
Quit attempts | Will be assessed by the participants in both groups by CO verification and self-administered online surveys.
  Will be assessed by the participants in both groups by CO verification and self-administered online surveys.
Smoking abstinence | At baseline, 4 weeks after start of intervention, and 1 week, 3 months and 6 months post-intervention
  Will be assessed by the amount of CO in a participant's breath using a portable carbon monoxide monitor, which is synced to the participants' smartphones and will ask participants to complete a brief smoking habit survey.

SECONDARY OUTCOMES:
Cigarette Dependence Scale (12 item) | Up to 6 months post-intervention
  This outcome will be assessed by the participants completing self-administered online survey that includes 12 questions.
Secondary measures that may contribute to smoking | At baseline, 1 week, 3 months and 6 months post-intervention
  Will include measures such as, anxiety and depression, physical activity, and pain. Will be assessed by the participants in both groups by self-administered online surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Ce Shang, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu